CLINICAL TRIAL: NCT00139568
Title: An Evaluation of the Efficacy and Safety of Tegaserod 6 mg Bid Given Orally to Chinese Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919E2308
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Constipation
Keywords: Chronic constipation; 5-HT,5-HT4,; functional GI; China; tegaserod
MeSH Terms: conditions — Constipation | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Tegaserod is an aminoguanidine indole compound and a member of a new class of 5-hydroxytryptamine (5-HT) agonists. Activation of 5-HT4 receptors triggers the release of neurotransmitters from the enteric nerves which in turn stimulate contractility and peristalsis. This study will investigate the efficacy and safety of tegaserod against chronic constipation in a Chinese population of adult men and women

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* History of constipation for at least 6 months prior to screening
* Normal bowel evaluation performed within the past 5 years

Exclusion Criteria:

* Most bothersome symptom in last 6 months is abdominal pain/discomfort
* Whose chronic constipation is thought to be a result of bowel surgery, gynecological surgery, neurologic disorder, systemic sclerosis, amyloidosis, scleroderma, myotonic dystrophy
* Insulin dependent diabetes
* Evidence of cathartic colon or laxative abuse

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-02; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of complete spontaneous bowel movements (CSBM) per week

SECONDARY OUTCOMES:
Response rate for CSBM during the first 4 weeks of treatment
Patients' daily assessment of bowel habits
Patients' weekly assessment of constipation symptoms
Satisfactory relief of CC symptoms
PAC-QoL questionnaire
PPSM questionnaire
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Basel, Switzerland
Locations (1):
- Novartis, Basel, Switzerland